CLINICAL TRIAL: NCT02194244
Title: A Randomized, Open-Label, Four Period, Four-Treatment Crossover Study to Investigate the Comparative Bioavailability of Film-Coated Tablet and Granule Formulations of RG1662 Under Fed and Fasted Conditions in Healthy Volunteers
Brief Title: Comparative Bioavailability Study of Film-coated Tablet and Granule Formulations of RG1662
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: WP28978; 2014-001762-97 (EudraCT Number)
Record Dates: First submitted 2014-07-08; First posted 2014-07-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (4):
- Granules Fasted (Experimental)
  Interventions: Drug: RG1662 granules
- Granules Fed (Experimental)
  Interventions: Drug: RG1662 granules
- Tablet Fasted (Active Comparator)
  Interventions: Drug: RG1662 tablet
- Tablet Fed (Active Comparator)
  Interventions: Drug: RG1662 tablet

INTERVENTIONS:
Drug: RG1662 granules — Single dose, oral administration of RG1662 immediate release granules
  Arms: Granules Fasted; Granules Fed
Drug: RG1662 tablet — Single dose, oral administration of film-coated RG1662 immediate release tablet
  Arms: Tablet Fasted; Tablet Fed

SUMMARY:
This study will compare the pharmacokinetic performance of film-coated tablet and granule formulations of RG1662 under fed and fasted conditions in healthy volunteers. A randomized, four-period, four-treatment crossover design is used. In each period, each volunteer will receive a single oral dose of the tablet or granule formulation either with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18 to 60 years of age, inclusive

Exclusion Criteria:

* A history of epilepsy, convulsions or significant head injury
* Any other clinically relevant abnormalities, concomitant diseases or ongoing medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Granules Fed (test): RG1662 plasma exposure, area under the concentration-time curve | Up to 9 weeks
Granules Fasted (test): RG1662 plasma exposure, area under the concentration-time curve | Up to 9 weeks
Tablet Fed (reference): RG1662 plasma exposure, area under the concentration-time curve | Up to 9 weeks
Tablet Fasted (reference): RG1662 plasma exposure, area under the concentration-time curve | Up to 9 weeks

SECONDARY OUTCOMES:
Tablet formulation: RG1662 plasma exposure ratio between fed (test) and fasted (reference) conditions, estimated from area under the concentration-time curve measurements | Up to 9 weeks
Granule formulation: RG1662 plasma exposure ratio between fed (test) and fasted (reference) conditions, estimated from area under the concentration-time curve measurements | Up to 9 weeks
Palatability of the granule formulation, as assessed by questionnaire | Day 1, Day 3 in granule administration periods
Safety: Incidence of adverse events with either formulation | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom